CLINICAL TRIAL: NCT03499223
Title: A Phase 2, Randomised, Single-masked, Active-controlled, Multicentre Study to Evaluate the Efficacy and Safety of Intravitreal THR-317 Administered in Combination With Ranibizumab, for the Treatment of Diabetic Macular Oedema (DME)
Brief Title: A Study to Evaluate THR-317 and Ranibizumab Combination Treatment for Diabetic Macular Oedema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxurion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THR-317-002; 2017-003897-15 (EudraCT Number)
Record Dates: First submitted 2018-04-04; First posted 2018-04-17 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Macular Edema | interventions — Ranibizumab; TB-403; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ranibizumab + THR-317 (Experimental): Subjects will receive intravitreal ranibizumab in combination with THR-317
  Interventions: Drug: Ranibizumab 0.5mg; Drug: THR-317 8mg
- Sham + ranibizumab (Active Comparator): Subjects will receive a sham injection in combination with intravitreal ranibizumab
  Interventions: Drug: Ranibizumab 0.5mg; Drug: Sham injection

INTERVENTIONS:
Drug: Ranibizumab 0.5mg — 3 intravitreal injections of ranibizumab 0.5mg, approximately 1 month apart
  Other Names: Lucentis®
Drug: THR-317 8mg — 3 intravitreal injections of THR-317 8mg, approximately 1 month apart
  Arms: Ranibizumab + THR-317
Drug: Sham injection — 3 sham injections, approximately 1 month apart. No actual injections. No medication is used.
  Arms: Sham + ranibizumab

SUMMARY:
This study is conducted to evaluate the safety of intravitreal THR-317 administered in combination with ranibizumab, and to assess the efficacy of the combination treatment in improving best-corrected visual acuity (BCVA) and reducing central subfield thickness (CST), in subjects with central-involved diabetic macular oedema (CI-DME).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Type 1 or type 2 Diabetes Mellitus
* CI-DME with central subfield thickness of ≥ 320μm on Spectralis® SD-OCT or ≥ 305μm on non Spectralis SD-OCT, in the study eye
* Anti-vascular endothelial growth factor (anti-VEGF) treatment naïve study eye, or poor or no response to prior treatment with ranibizumab in the study eye
* Reduced vision primarily due to DME, with BCVA ≤ 72 and ≥ 23 ETDRS letter score (≤ 20/40 and ≥ 20/320 Snellen equivalent) in the study eye
* Non-proliferative diabetic retinopathy of any stage in the study eye
* Written informed consent obtained from the subject prior to screening procedures

Exclusion Criteria:

* Concurrent disease in the study eye, other than CI-DME, that could compromise BCVA, require medical or surgical intervention during the study period or could confound interpretation of the results
* Previous confounding treatments / procedures, or their planned / expected use during the study period for up to 30 days after the last administration of study treatment
* Any active ocular / intraocular infection or inflammation in either eye
* Aphakic study eye
* Poorly controlled Diabetes Mellitus
* Uncontrolled hypertension
* Pregnant or lactating female, or female of child-bearing potential not utilising an adequate form of contraception, or male of reproductive potential not utilising contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BCVA | At Day 84 (Month 3)

SECONDARY OUTCOMES:
Incidence of systemic and ocular adverse events including serious adverse events | From Day 0 to Day 140
Change from baseline in BCVA, by study visit | From Day 0 to Day 140
Change from baseline in CST, based on spectral domain optical coherence tomography (SD-OCT), as assessed by the central reading centre, by study visit | From Screening to Day 140
Withdrawal from repeat study treatment and reason for withdrawal | At Day 28 and at Day 56
  Number of subjects meeting withdrawal criteria from repeat study treatment

CONTACTS AND LOCATIONS:
Locations (37):
- Belgium (2):
  - CHU Brugmann, Brussels
  - UZ Leuven, Leuven
- France (10):
  - Centre Rétine Gallien, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Dijon, Dijon
  - Hôpital Privé La Louvière, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Nice, Hôpital Pasteur, Nice
  - Centre Ophtalmologique de l'Odéon, Paris
  - Hôpital Lariboisière, Paris
  - Centre Ophtalmologique Maison Rouge, Strasbourg
- Germany (6):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Philipps-Universität Marburg, Marburg
- Slovakia (5):
  - Univerzitná nemocnica Bratislava, Nemocnica Ružinov, Bratislava
  - Univerzitná nemocnica Bratislava, Nemocnica Sv. Cyrila a Metoda, Bratislava
  - Nemocnica Poprad, a.s., Poprad
  - Fakultná nemocnica Trenčín, Trenčín
  - Fakultná nemocnica s polikliniku Žilina, Žilina
- Spain (8):
  - Centro Médico Téknon, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital general de Cataluña, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Vissum Madrid, Madrid
  - Hospital General Universitario de Valencia, Valencia
  - Oftalvist IMED Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- RétinElysée, Lausanne, Switzerland
- United Kingdom (5):
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland